CLINICAL TRIAL: NCT01326013
Title: A Two-Arm, Multi-Centre Clinical Evaluation of the xTAG Gastrointestinal Pathogen Panel (xTAG GPP) in Patients With Signs and Symptoms of Infectious Colitis and Gastroenteritis
Brief Title: A Two-Arm, Multi-Centre Clinical Evaluation of the xTAG Gastrointestinal Pathogen Panel
Status: Completed | Type: Observational
Sponsor: Luminex Molecular Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: TDP-736-189
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Infectious; Colitis; Gastroenteritis
Keywords: Stool; Feces; Gastrointestinal; Pathogen; Panel; xTAG GPP; Infectious colitis; Gastroenteritis; Detection
MeSH Terms: conditions — Communicable Diseases; Colitis; Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blinded, Prospective Arm: Diagnostic accuracy for higher prevalence targets will be evaluated in prospectively collected, anonymized, leftover, stool specimens.
- Blinded, Pre-selected Arm: For targets that exhibit lower prevalence rates in the intended use population, banked, pre-selected, positive clinical specimens will be tested.

SUMMARY:
The xTAG Gastrointestinal Pathogen Panel (xTAG GPP) is a PCR-based assay to detect the presence or absence of gastrointestinal (GI) pathogens from human stool specimens.

The objective of this study is to establish diagnostic accuracy of the xTAG GPP.

DETAILED DESCRIPTION:
The xTAG GPP assay is a qualitative nucleic acid multiplex test intended to simultaneously detect and identify bacterial (and toxins), viral, and parasitic pathogens extracted from human stool specimens collected from patients with signs and symptoms of infectious colitis or gastroenteritis.

The objective of this study is to establish the diagnostic accuracy of xTAG GPP through a multi-site, method comparison study on prospectively collected, left-over, and anonymized stool specimens. The prospective sample set will also be supplemented with pre-selected archived left-over specimens (for low prevalence targets only). Diagnostic accuracy will be expressed in terms of clinical sensitivity and specificity for each target.

ELIGIBILITY:
Inclusion Criteria:

* The specimen is stool.
* The specimen is from a pediatric or adult, male or female subject who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinic or resident of a long-term care facility.
* The specimen is from a patient exhibiting clinical signs and symptoms of infectious colitis or gastroenteritis.

Exclusion Criteria:

* The specimen is a preserved stool, stool in Cary-Blair media or rectal swab.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical specimens collected from patients with signs and symptoms of infectious colitis or gastroenteritis who are either hospitalized, admitted to emergency departments or visiting outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 1534 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Liu, Ph.D, Study Director — Luminex Molecular Diagnostics; Tony Mazzulli, M.D., F.R.C.P.(C), FACP, Principal Investigator — MOUNT SINAI HOSPITAL; Robert C. Fader, Ph.D, Principal Investigator — Scott and White Hospital & Clinic; James Mahony, Ph.D, FCCM, FAAM, Principal Investigator — St. Joseph's Hospital; Yi-Wei Tang, M.D., Ph.D, Principal Investigator — Vanderbilt University Medical Centre; Richard Buller, Ph.D., D(ABMM), Principal Investigator — St. Louis Children's Hospital; Donna M. Wolk, Ph.D., D.(ABMM), Principal Investigator — University of Arizona
Locations (6):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - St. Louis Children's Hospital, St Louis, Missouri
  - Vanderbilt University Medical Centre, Nashville, Tennessee
  - Scott and White Memorial Hospital, Temple, Texas
- Canada (2):
  - St. Joseph's Hospital, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario